CLINICAL TRIAL: NCT03475381
Title: Real-life Follow-up of Cystic Fibrosis Patients Treated With Ivacaftor+Lumacaftor (Orkambi*)
Acronym: ORKAMBI
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Effi-Stat (Other); Societe Francaise de la Mucoviscidose (Other); URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Other Study IDs: NI17043HLJ
Record Dates: First submitted 2018-01-04; First posted 2018-03-23 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Cystic Fibrosis
Keywords: Cystic Fibrosis; ivacaftor; lumacaftor
MeSH Terms: conditions — Cystic Fibrosis | interventions — lumacaftor, ivacaftor drug combination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Orkambi treated patients: All patients with CF who started ivacaftor+lumacaftor outside of a clinical trial between January 22nd 2016 and January 22nd 2017.
  Interventions: Drug: Ivacaftor+lumacaftor

INTERVENTIONS:
Drug: Ivacaftor+lumacaftor — 1 year follow-up after initiation of ivacaftor+lumacaftor
  Other Names: Orkambi

SUMMARY:
The purpose of the study is to examine the real-life safety and effectiveness of the novel combination ivacaftor+lumacaftor in eligible patients with cystic fibrosis (CF). All patients with CF were eligible if they were 12 years and older, started ivacaftor+lumacaftor outside of a clinical trial between December 15th 2017 and December 15th 2018 in an accredited CF center in France. Patient followed-up is based on standardized recommendation of the French Cystic Fibrosis Society. Each patient is followed 1 year.

DETAILED DESCRIPTION:
Each patient is followed one year with visits at months 1, 3, 6 and 12.

At each visit, the following data are recorded:

* Treatment discontinuation or not. If the treatment was discontinued, reasons for discontinuation
* Adverse effects
* Lung function (spirometry)
* Body mass index
* Pulmonary exacerbations (intravenous antibiotics)
* Sputum microbiology
* Liver enzymes are measured at each visit

At the initial and 12 visits, a yearly CF examination is proposed to the patients:

* Blood tests
* Chest CT scans
* Body plethysmography

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 12 years or older.
* Patient with Cystic Fibrosis with presence of two mutations DF508 in the CFTR gene
* Patient treated with ivacaftor+lumacaftor (Orkambi)

Exclusion Criteria:

* Refusal to participate in the study
* Start of Orkambi as part of a clinical trial

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patient with Cystic Fibrosis with presence of two mutations DF508 in the CFTR gene and treated by Orkambi in usual care
Sampling Method: Non-Probability Sample
Enrollment: 852 (Actual)
Dates: Start 2016-01-22 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Rates of treatment discontinuation | 1 year
Timing of treatment discontinuation | 1 year
Causes of treatment discontinuation | 1 year

SECONDARY OUTCOMES:
Forced expiratory volume in 1 sec (FEV1) | 1 year
  to evaluate lung function
Forced vital capacity (FVC) | 1 year
  to evaluate lung function
Body mass index | 1 year
  Nutritional status
Pulmonary exacerbations | 1 year
  Intravenous antibiotic courses
Chloride concentration | 1 year
  Sweat test before and during treatment

CONTACTS AND LOCATIONS:
Overall Officials: Pierre-Regis BURGEL, MD, PhD, Principal Investigator — Hôpitaux Universitaire Paris Centre, AP-HP
Locations (1):
- Adult CF center, Service de Pneumologie, Cochin Hospital, Paris, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Burgel PR, Munck A, Durieu I, Chiron R, Mely L, Prevotat A, Murris-Espin M, Porzio M, Abely M, Reix P, Marguet C, Macey J, Sermet-Gaudelus I, Corvol H, Bui S, Lemonnier L, Dehillotte C, Da Silva J, Paillasseur JL, Hubert D; French Cystic Fibrosis Reference Network Study Group. Real-Life Safety and Effectiveness of Lumacaftor-Ivacaftor in Patients with Cystic Fibrosis. Am J Respir Crit Care Med. 2020 Jan 15;201(2):188-197. doi: 10.1164/rccm.201906-1227OC. PMID 31601120